CLINICAL TRIAL: NCT01840787
Title: A Pilot Study on the Use of a Sensory Panel to Assess Comfort Between Three Different Contact Lenses
Acronym: NAISMITH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: 18801
Record Dates: First submitted 2013-04-19; First posted 2013-04-26 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contralateral lens comfort comparisons (Experimental): Subjects will be randomized into receiving balafilcon A (8.3), or balafilcon A (8.6), or senofilcon A in one eye, and balafilcon A (8.3), or balafilcon A (8.6), or senofilcon A in the other eye.
  Interventions: Device: balafilcon A (8.6); Device: balafilcon A (8.3); Device: senofilcon A

INTERVENTIONS:
Device: balafilcon A (8.6) — To be worn for 8 hours in one eye, and its comfort compared to another lens on another eye.
  Other Names: Bausch & Lomb PureVision 8.6
Device: balafilcon A (8.3) — To be worn for 8 hours in one eye, and its comfort compared to another lens on another eye.
  Other Names: Bausch & Lomb PureVision 8.3
Device: senofilcon A — To be worn for 8 hours in one eye, and its comfort compared to another lens on another eye.
  Other Names: Johnson & Johnson Acuvue Oasys

SUMMARY:
As new contact lens products continue to be developed and improved, it's becoming harder for some individuals to tell whether one product is different from another. In addition, not everyone has the same level of sensitivity of their eyes, making it difficult for these judgments to be made. The purpose of this study is to explore the idea of using a pre-determined "expert panel" of individuals who are able to tell differences between contact lenses based on their comfort.

DETAILED DESCRIPTION:
As technology continues to advance, contact lenses and lens care products are becoming harder to differentiate. In addition, assessing comfort in clinical trials is complicated, with full-masking behind hard to achieve and the psychology of the participant having unknown impact on the results. While the development of a reliable system to assess comfort would be beneficial for the research and development of new products, the use of a "sensory panel" itself may also lead to a better understanding of the drivers of discomfort at the end of the day.

The objective of the study is to explore the use of a sensory panel, defined as individuals who have a good correlation between subjective and objective measures of discomfort, at rating the comfort of various contact lenses.

The hypothesis is that in the "discriminative" group, the matrix of paired comparisons (between lens dissimilarity) is related to the ranked comfort of the lenses, while for the "poorly discriminative" group, the matrix of the dissimilarities will be random. An additional hypothesis is that the "discriminative" group will be less random than the entire group.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Is an adapted soft contact lens wearer;
* Has a contact lens prescription between +4.00 to -6.00D;
* Has astigmatism <= 1.00D;
* Has vision of 20/40 or better in both eyes when wearing contact lenses

Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Has any known active ocular disease and/or infection;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Is pregnant, lactating or planning a pregnancy at the time of enrolment, determined verbally;
* Is aphakic;
* Has undergone refractive surgery;
* Is an employee of the Centre for Contact Lens Research;
* Has anisometropia of >=1.00D
* Has a difference in comfort of 20 (on a 0-100 scale) between eyes when not wearing contact lenses.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in eye comfort ratings | Prior to, and after lens insertion in the morning, and then again 8 hours later.

CONTACTS AND LOCATIONS:
Overall Officials: Trefford Simpson, DipOptom, Principal Investigator — University of Waterloo School of Optometry & Vision Science
Locations (1):
- Centre for Contact Lens Research, University of Waterloo School of Optometry & Vision Science, Waterloo, Ontario, Canada